CLINICAL TRIAL: NCT01110694
Title: Prospective Observation of Fibrosis in the Lung Clinical Endpoints (PROFILE_Brompton)Study
Brief Title: Prospective Observation of Fibrosis in the Lung Clinical Endpoints Study
Acronym: PROFILE
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry); University College, London (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: PROFILE_RBH_001; 10/H0720/12 (Other: Royal Free Hospital REC)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Idiopathic Non-specific Interstitial Pneumonitis
Keywords: Idiopathic pulmonary fibrosis; Interstitial lung disease; Prognosis; Biomarkers; Mortality; Acute exacerbations
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, bronchoalveolar lavage, surgical lung biopsy (when clinically indicated)
Oversight: Data Monitoring Committee: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a progressive scarring condition of the lungs the cause of which is unknown.There are currently no effective treatments for IPF and the condition tends to cause progressive disability and death with an average survival of 3.5 years from diagnosis. The condition is responsible for the deaths of 4000 people per year in the UK. At present the definite diagnosis of IPF rests on the identification of a specific pattern of fibrosis when a section of fibrotic lung tissue is examined under a microscope. Unfortunately, the process of obtaining a lung biopsy requires an operation and is not with out risk. The investigators hope to identify specific markers in the blood and lungs of patients with IPF that will enable the condition to be diagnosed without biopsy. Furthermore, the investigators hope to identify indicators(biomarkers) that will predict which patients have more aggressive and progressive disease and also to identify biomarkers that might be useful in identifying a response to treatment and might therefore be used in future clinical trials in IPF. As well as looking at markers in the blood and lungs the investigators also plan to assess the use of daily home lung function measurement and a computerised technique for analyzing lung sounds to see if these are investigations that are able to predict the development of worsening lung fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 with a diagnosis of definite or probable IPF or definite or probable fibrotic NSIP as defined by the ATS/ERS consensus classification

Exclusion Criteria:

* Patients with co-existent conditions known to be associated with the development of fibrotic lung disease will be excluded.
* This includes

  * connective tissue disease
  * suspected drug-induced lung disease
  * asbestosis or other asbestos related disease (pleural plaques, mesothelioma, asbestos pleural effusions)
  * granulomatous disease including sarcoidosis.
* Patients with an auto-immune profile considered diagnostic for a specific connective tissue disease will be excluded, even in the absence of systemic symptoms.
* Non-specific rises in auto antibodies e.g. rheumatoid factor, anti-nuclear antibody etc. will not be used to exclude individuals from the study.
* Patients with co-morbid disease that in the opinion of the investigators gives them an expected life expectancy of less than one year will be excluded from the study.
* Patients involved in clinical trials assessing novel IPF therapies will be excluded from enrolment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients refered to the Interstitial Lung Disease Unit of the Royal Brompton Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Biomarker discovery | 3 years
  Discover and validate novel biomarkers and gene expression profiles for use in subsequent clinical studies in patients with idiopathic pulmonary fibrosis.

SECONDARY OUTCOMES:
Study disease behaviour | 3 years
  Prospectively evaluate longitudinal disease behavior in patients with IPF and other fibrotic lung diseases of unknown cause with a view to developing composite clinical endpoints for subsequent use in clinical studies in patients with pulmonary fibrosis.
Differentiate IPF from NSIP | 3 years
  Identify differences in the pathogenetic mechanisms involved in the development of different types of fibrosis in patients with fibrotic lung disease of unknown cause.

CONTACTS AND LOCATIONS:
Overall Officials: Toby M Maher, MB PhD, Principal Investigator — Royal Brompton and Harefield Foundation NHS Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Background] Maher TM, Wells AU, Laurent GJ. Idiopathic pulmonary fibrosis: multiple causes and multiple mechanisms? Eur Respir J. 2007 Nov;30(5):835-9. doi: 10.1183/09031936.00069307. PMID 17978154
- [Background] Gribbin J, Hubbard RB, Le Jeune I, Smith CJ, West J, Tata LJ. Incidence and mortality of idiopathic pulmonary fibrosis and sarcoidosis in the UK. Thorax. 2006 Nov;61(11):980-5. doi: 10.1136/thx.2006.062836. Epub 2006 Jul 14. PMID 16844727
- [Background] Maher TM. The diagnosis of idiopathic pulmonary fibrosis and its complications. Expert Opin Med Diagn. 2008 Dec;2(12):1317-31. doi: 10.1517/17530050802549484. PMID 23496780
- [Background] Hubbard R, Johnston I, Britton J. Survival in patients with cryptogenic fibrosing alveolitis: a population-based cohort study. Chest. 1998 Feb;113(2):396-400. doi: 10.1378/chest.113.2.396. PMID 9498958
- [Background] Moeller A, Gilpin SE, Ask K, Cox G, Cook D, Gauldie J, Margetts PJ, Farkas L, Dobranowski J, Boylan C, O'Byrne PM, Strieter RM, Kolb M. Circulating fibrocytes are an indicator of poor prognosis in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2009 Apr 1;179(7):588-94. doi: 10.1164/rccm.200810-1534OC. Epub 2009 Jan 16. PMID 19151190
- [Background] Maher TM. Understanding nonspecific interstitial pneumonia: the need for a diagnostic gold standard. Am J Respir Crit Care Med. 2009 Feb 1;179(3):255-6; author reply 256. doi: 10.1164/ajrccm.179.3.255. No abstract available. PMID 19158329
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Maher TM, Oballa E, Simpson JK, Porte J, Habgood A, Fahy WA, Flynn A, Molyneaux PL, Braybrooke R, Divyateja H, Parfrey H, Rassl D, Russell AM, Saini G, Renzoni EA, Duggan AM, Hubbard R, Wells AU, Lukey PT, Marshall RP, Jenkins RG. An epithelial biomarker signature for idiopathic pulmonary fibrosis: an analysis from the multicentre PROFILE cohort study. Lancet Respir Med. 2017 Dec;5(12):946-955. doi: 10.1016/S2213-2600(17)30430-7. Epub 2017 Nov 14. PMID 29150411
- [Derived] Jenkins RG, Simpson JK, Saini G, Bentley JH, Russell AM, Braybrooke R, Molyneaux PL, McKeever TM, Wells AU, Flynn A, Hubbard RB, Leeming DJ, Marshall RP, Karsdal MA, Lukey PT, Maher TM. Longitudinal change in collagen degradation biomarkers in idiopathic pulmonary fibrosis: an analysis from the prospective, multicentre PROFILE study. Lancet Respir Med. 2015 Jun;3(6):462-72. doi: 10.1016/S2213-2600(15)00048-X. Epub 2015 Mar 12. PMID 25770676